CLINICAL TRIAL: NCT05594238
Title: Leveraging Virtual Care Strategies to Improve Access and Treatment for Individuals With Alcohol Use Disorders (AUD)
Brief Title: Leveraging Virtual Care Strategies to Improve Access and Treatment for Individuals With Alcohol Use Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Erin Bonar, Associate Professor, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00210546; R01AA029808 (NIH)
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: Telehealth
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants are first randomly assigned to two interventions: either Telephone Engagement or Portal Engagement. Participants who do not meet the criteria for response at the post-test will be re-randomized into either enhanced first stage or a Telehealth MI-CBT program.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A (Active Comparator): First stage intervention: Telephone engagement Second stage intervention: Telehealth Motivational Interviewing-Cognitive Behavioral Therapy (MI-CBT program)
  Interventions: Behavioral: Telephone Engagement; Behavioral: MI-CBT
- Arm B (Active Comparator): First stage intervention: Telephone engagement Second stage intervention: Enhanced Telephone engagement
  Interventions: Behavioral: Telephone Engagement
- Arm C (Active Comparator): First stage intervention: Telephone engagement Second stage intervention: Not Applicable (NA), proceed directly to follow up
  Interventions: Behavioral: Telephone Engagement
- Arm D (Active Comparator): First stage intervention: Portal Engagement Second stage intervention: NA, proceed directly to follow up
  Interventions: Behavioral: Portal Engagement
- Arm E (Active Comparator): First stage intervention: Portal Engagement Second stage intervention: Enhanced Portal Engagement
  Interventions: Behavioral: Portal Engagement
- Arm F (Active Comparator): First stage intervention: Portal Engagement Second stage intervention: Telehealth MI-CBT program
  Interventions: Behavioral: Portal Engagement; Behavioral: MI-CBT

INTERVENTIONS:
Behavioral: Telephone Engagement — Brief phone session with a study counselor.
  Arms: Arm A; Arm B; Arm C
Behavioral: Portal Engagement — Access to a virtual portal where participant messages with study counselors.
  Arms: Arm D; Arm E; Arm F
Behavioral: MI-CBT — 8 one-on-one sessions done over the phone or video chat with a study counselor
  Arms: Arm A; Arm F

SUMMARY:
The purpose of this research study is to test new technology-driven programs to see if they might help people manage their health and health behaviors related to alcohol use and well-being. The programs focus on getting to know what's important to participants, reviewing or setting goals, and using different skills and behaviors to manage health. The study will help researchers learn about ways to deliver health information in a way that is useful and interesting.

ELIGIBILITY:
Inclusion Criteria:

* AUD
* past month heavy alcohol use
* internet access
* phone access
* able to provide informed consent

Exclusion Criteria:

* inability to speak or understand English
* conditions precluding informed consent or understanding of intervention or assessment content
* recent AUD treatment
* history of or at risk for complex alcohol withdrawal
* involvement in another ongoing study for alcohol/mental health/substance use treatment
* current cancer diagnosis/ currently receiving cancer treatment (other than skin cancers)
* PI discretion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
AUD Treatment Initiation | 4-months post-enrollment
  % of patients who initiate psychotherapy treatment
AUD Treatment Engagement | 4-months post-enrollment
  % of patients who attend at least 2 psychotherapy treatment sessions
Alcohol consumption days | 4-months post-enrollment
  % of days of alcohol consumption as measured by the Timeline Follow Back Interview
Alcohol consumption days | 8-months post-enrollment
  % of days of alcohol consumption as measured by the Timeline Follow Back Interview
Alcohol consumption days | 12-months post-enrollment
  % of days of alcohol consumption as measured by the Timeline Follow Back Interview
Heavy drinking days | 4-months post-enrollment
  % of days of heavy drinking as measured by the Timeline Follow Back Interview
Heavy drinking days | 8-months post-enrollment
  % of days of heavy drinking as measured by the Timeline Follow Back Interview
Heavy drinking days | 12-months post-enrollment
  % of days of heavy drinking as measured by the Timeline Follow Back Interview

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Bonar, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with sponsor requirements, de-identified data will be shared with the NIAAA Data Repository, if participants agree.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Bonar EE, Kidwell K, Chapman L, Walton MA, Zheng K, Bourque C, Manderachia D, Robinson OE, Eissa AA, Dailey SE, Dolecki F Jr, Teasdale OD, NanCoff A, Chizek EE, Tyner TS, Miller AL, Lin LA. Telehealth engagement and treatment strategies for adults living with alcohol use disorder: A sequential multiple assignment randomized trial protocol. Contemp Clin Trials. 2025 Sep;156:108003. doi: 10.1016/j.cct.2025.108003. Epub 2025 Jul 9. PMID 40645371